CLINICAL TRIAL: NCT07346014
Title: Triple Chronotherapy + Transdiagnostic Sleep and Circadian Intervention (TSC+) for Suicidal Young Adults
Brief Title: Sleep and Circadian Interventions for College Students at High Risk of Suicide
Acronym: REST-UP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Tina R Goldstein, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY25060093; BSG-0-204-24 (Other Grant/Funding Number: American Foundation for Suicide Prevention)
Record Dates: First submitted 2026-01-06; First posted 2026-01-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disturbance; Sleep; Depression; Suicide
Keywords: sleep disturbance; suicide; triple chronotherapy
MeSH Terms: conditions — Parasomnias; Depression; Suicide | interventions — Thrombin Time

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sleep Feedback + Psychoeducation (Experimental): Participants receive an actigraphy watch to track their sleep and activity levels and complete a daily sleep diary; sleep feedback graphs show participants their actigraphy watch and sleep diary data on demand.
  Interventions: Behavioral: Sleep Feedback + Psychoeducation
- Transdiagnostic Sleep and Circadian Intervention + Bright Light (TSC+) (Experimental): Participants will attend 6-8 TSC sessions of a manualized sleep intervention with a Sleep therapist, delivered in person or videoconference. Participants will also wear bright light glasses (up to 60 minutes) in the morning and blue light blocking glasses in the evening throughout the intervention.
  Additionally, participants receive an actigraphy watch to track their sleep and activity levels and complete a daily sleep diary; sleep feedback graphs show participants their actigraphy watch and sleep diary data on demand.
  Interventions: Behavioral: Sleep Feedback + Psychoeducation; Behavioral: Transdiagnostic Sleep and Circadian Intervention + Bright Light (TSC+)
- Triple Chronotherapy + Transdiagnostic Sleep and Circadian Intervention + Bright Light (TSC+) (Experimental): TCT+ Participants receive a four-day intervention, beginning with an approximately 33-hour total sleep deprivation period, followed by 3-days of sleep phase advancement and daily bright light therapy (up to sixty minutes) in the morning and blue light blocking glasses (up to one hour before bedtime) in the evening, in a sleep lab.
  TSC+ Participants will also attend 6-8 TSC sessions of a manualized sleep intervention with a Sleep therapist, delivered in person or videoconference. Participants will continue to wear bright light glasses (up to sixty minutes daily) in the morning and blue light blocking glasses (up to one hour before bedtime) in the evening throughout the intervention.
  SF Participants receive an actigraphy watch to track their sleep and activity levels and complete a daily sleep diary; sleep feedback graphs show participants their actigraphy watch and sleep diary data on demand.
  Interventions: Behavioral: Sleep Feedback + Psychoeducation; Behavioral: Transdiagnostic Sleep and Circadian Intervention + Bright Light (TSC+); Behavioral: Triple Chronotherapy (TCT+)

INTERVENTIONS:
Behavioral: Sleep Feedback + Psychoeducation — Participants are provided with an actigraphy watch that is used to monitor their sleep and activity throughout the day and complete a sleep diary daily. Along with wearing the watch they also will be provided access to their actigraphy and sleep diary graphs that document their data on demand via smartphone link.
Behavioral: Transdiagnostic Sleep and Circadian Intervention + Bright Light (TSC+) — Behavioral: TSC+
  • This intervention includes participants attending 6-8 sessions of a manualized sleep intervention with a Sleep Therapist, delivered in person or videoconference, as well as daily bright light therapy (up to one hour daily) and blue light blocking glasses (up to one hour before bedtime)
  Arms: Transdiagnostic Sleep and Circadian Intervention + Bright Light (TSC+); Triple Chronotherapy + Transdiagnostic Sleep and Circadian Intervention + Bright Light (TSC+)
Behavioral: Triple Chronotherapy (TCT+) — Behavioral: TCT+
  • One night of total sleep deprivation followed by three nights of sleep phase advancement in the sleep lab, daily bright light therapy (up to one hour daily) and blue light blocking glasses (up to one hour before bedtime), in a sleep lab.
  Arms: Triple Chronotherapy + Transdiagnostic Sleep and Circadian Intervention + Bright Light (TSC+)

SUMMARY:
The purpose of this study is to examine the extent to which delivering sleep and circadian focused interventions in addition to evidenced based psychiatric care for depression and suicide risk may contribute to decreasing suicide risk among high risk young adults. Investigators will evaluate three interventions targeting sleep in acutely suicidal college students enrolled in intensive outpatient treatment. Participants will be randomly assigned to one of three intervention groups:

1. Triple Chronotherapy (TCT)+ Transdiagnostic Sleep and Circadian Intervention (TSC)
2. Transdiagnostic Sleep and Circadian Intervention (TSC)
3. Sleep Feedback (SF) Participants will be followed for 6 months with primary outcome domains of suicidal thoughts and behaviors and depression evaluated by blinded clinicians at short (Days 1-4 of intervention), medium (2 months) and long (6 month) term intervals.

DETAILED DESCRIPTION:
Suicide is currently the second leading cause of death among college students, and suicidal thoughts and behaviors (STBs) in this group have increased substantially in recent years. Indeed, young adulthood represents a particularly high-risk period for onset of psychiatric disorders associated with STBs, including depression, anxiety, and substance use disorder. There is a pressing need for efficacious treatments for suicidal college students that yield fast-acting and sustained effects in order to minimize disruption to young adults' developmental trajectories. While efficacious treatments exist to decrease suicide risk, effects generally take months. Interventions that rapidly improve suicidality are thus urgently needed. Triple chronotherapy (TCT) is a candidate, as two open studies documented dramatic reductions in suicidality. TCT is a 4-5 day intervention that involves one day and night of sleep deprivation, followed by 4 nights of sleep advance of bed/waketimes combined with morning bright light therapy (presumed to both advance the circadian rhythm and improve mood). Randomized control trials indicate that TCT rapidly improves depression, though suicide-specific randomized control trials have not been conducted to date. The investigators will thus propose to examine TCT as a means to rapidly reduce suicidality, but to also pair this with a multidimensional sleep health intervention (i.e., the Transdiagnostic Sleep and Circadian Intervention, TSC) to test whether this will help sustain improvements. Investigators assert that a "TCT+" package that includes TCT (4-day protocol) followed by TSC+ (6-8 outpatient sessions) holds promise to safely and non-invasively yield rapid and sustained improvement in depression and STBs among suicidal college students. This study is a 3-arm RCT comparing TCT+ vs TSC+ Alone vs Sleep Feedback (Ctrl) in 90 acutely suicidal college students, ages 18-25 years, reporting sleep difficulties and receiving Intensive Outpatient Program (IOP) treatment. The investigators will examine trajectories of depression and suicidality over short- (i.e., 4 days), medium- (i.e., 2 months), and long-term (i.e., 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled or planning to enroll in treatment at COSTAR Intensive Outpatient Program
* English language fluency and literacy sufficient to engage in study protocol
* Suicidal ideation or suicide attempt in past month
* Clinically significant sleep disturbance, operationalized as Pittsburgh Sleep Quality Index global PSQI score >= 7, and/or delayed bedtimes (>midnight), and/or >2 hours in sleep timing variability

Exclusion Criteria:

* Non-affective psychosis per electronic health record (EHR) review and/or baseline clinical assessment, or symptom severity or psychosocial functioning impairments that preclude participation
* Contraindications for either sleep deprivation or bright light therapy (e.g., bipolar disorder; seizure disorder; photosensitizing medication)
* Intellectual disability precluding comprehension of study procedures
* Evidence of untreated obstructive sleep apnea and/or restless legs syndrome
* Life-threatening medical condition requiring immediate treatment (such as cancer; end stage disease)
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Suicidal Thoughts and Behaviors via CSSRS | (short term) Intervention Days 1-4
  Columbia Suicide Severity Rating Scale, administered via clinician on Intervention Days 1-4. Range of 0-5, higher values represent higher severity/intensity
Suicidal Thoughts and Behaviors via CSSRS | (medium term) 2 month follow up
  Columbia Suicide Severity Rating Scale, administered via clinician at 2 month follow up assessment. Range of 0-5, higher values represent higher severity/intensity
Suicidal Thoughts and Behaviors via CSSRS | (long term) 6 month follow up
  Columbia Suicide Severity Rating Scale, administered via clinician at 6 month follow up assessment. Range of 0-5, higher values represent higher severity/intensity
Suicidal Thoughts and Behaviors via LIFE SI/SIB scale | (medium term) 2mo follow up
  The Longitudinal Interval Follow-Up Evaluation (LIFE) Self Injurious/Suicidal Behaviors Measure, administered by clinician at the 2-month assessment (LIFE SI/SIB Range 0-5, higher number indicates greater lethality)
Suicidal Thoughts and Behaviors via LIFE SI/SIB scale | (long term) 6mo follow up
  The Longitudinal Interval Follow-Up Evaluation (LIFE) Self Injurious/Suicidal Behaviors Measure, administered by clinician at the 6-month assessment (LIFE SI/SIB Range 0-5, higher number indicates greater lethality)
Depression via KSADS Depression Rating Scale | (short term) Intervention Days 1-4
  The Kiddie Schedule for Affective Disorders and Schizophrenia-Depression Rating Scale, administered via clinician at Intervention Days 1-4. (KDRS Range 0-64 with higher scores indicating greater severity)
Depression via KSADS Depression Rating Scale | (medium term) 2mo follow up
  The Kiddie Schedule for Affective Disorders and Schizophrenia-Depression Rating Scale, administered via clinician at 2 month follow up. (KDRS Range 0-64 with higher scores indicating greater severity)
Depression via KSADS Depression Rating Scale | (long term) 6mo follow up
  The Kiddie Schedule for Affective Disorders and Schizophrenia-Depression Rating Scale, administered via clinician at 6 month follow up. (KDRS Range 0-64 with higher scores indicating greater severity)
Depression via LIFE PSR | (medium term) 2mo follow up
  The Longitudinal Interval Follow-Up Evaluation (LIFE) Psychiatric Status Ratings, administered by clinician at the 2 month assessment (PSR; Range 1-6, higher numbers indicate greater severity)
Depression via LIFE PSR | (long term) 6mo follow up
  The Longitudinal Interval Follow-Up Evaluation (LIFE) Psychiatric Status Ratings, administered by clinician at the 6 month assessment (PSR Range 1-6, higher numbers indicate greater severity)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Goldstein, PhD, Principal Investigator — University of Pittsburgh; Peter Franzen, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Hospital/University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No